CLINICAL TRIAL: NCT04486079
Title: Preoperative Carbohydrate Loading in Bariatric Surgery - Randomized Clinical Trail
Brief Title: Preoperative Carbohydrate Loading in Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PreOpxBariatric
Record Dates: First submitted 2020-07-12; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Obesity, Morbid
Keywords: bariatric surgery; carbohydrate loading; insulin resistance
MeSH Terms: conditions — Obesity, Morbid; Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohyrate loading (Experimental): Group A will receive 400ml of the carbohydrate rich drink, Nutricia preOp 2 hours before operation. This is the intervention group.
  Interventions: Dietary Supplement: Nutricia PreOp
- Fasting (No Intervention): Group B will be prepared before the operation with a 24-hour fasting. This is the current clinical standard.

INTERVENTIONS:
Dietary Supplement: Nutricia PreOp — A clear, non-carbonated lemon-flavored, iso-osmolar carbohydrate drink for preoperative surgical patients. Used in studies supporting the Enhanced Recovery After Surgery (ERAS) Society Consensus Guidelines.
  Arms: Carbohyrate loading

SUMMARY:
The aim of this study is to perform a randomized non-blinded clinical trial to assess influence of preoperative carbohydrates loading in patients undergoing bariatric surgery measured by changes in the course of the postoperative period, changes in body composition and changes in insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* Obtaining written and informed patient consent.
* No medical contraindications to perform a bariatric operation
* No contraindications for the use of a rich carbohydrate drink

Exclusion Criteria:

* No consent to participate in the study
* Age under 18 years
* The intolerance of the carbohydrate drink used in the test
* The contraindications to perform bioimpedance measurements of body composition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
QoR40 score | 1st postoperatie day
  Quality of recovery after surgery will be assessed by the QoR40 survey Full scale title: Quality of Recovery 40-item questionnaires range from 40 (extremely poor. quality of recovery) to 200 (excellent quality of recovery)

SECONDARY OUTCOMES:
HOMA-IR | first assay one month before the operation, the second assay on the first postoperative day
  changes in insulin resistance will be assessed with HOMA index (Homeostatic Model Assessment for Insulin Resistance)
Body composition | first assay one month before the operation, the second assay on the first postoperative day
  changes in body composition will be assessed by electric bioimpedance method
Length of hospital stay | From the time of hospital admission following surgery, until the time of hospital discharge; assessed from day of hospital admision up to 30 days
  length of stay record in hours

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Wilczyński, Principal Investigator — General Surgery Resident, PhD Fellow, Teaching Assistant
Locations (1):
- Department of General, Endocrine and Transplant Surgery Medical University of Gdańsk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Medical University of Gdańsk will be the owner of data

REFERENCES:
- [Result] Knight P, Chou J, Dusseljee M, Verseman S, Elian A. Effective reduction in stress induced postoperative hyperglycemia in bariatric surgery by better carb loading. Am J Surg. 2020 Mar;219(3):396-398. doi: 10.1016/j.amjsurg.2019.10.042. Epub 2019 Nov 9. PMID 31757437
- [Result] Grant MC, Gibbons MM, Ko CY, Wick EC, Cannesson M, Scott MJ, McEvoy MD, King AB, Wu CL. Evidence Review Conducted for the Agency for Healthcare Research and Quality Safety Program for Improving Surgical Care and Recovery: Focus on Anesthesiology for Bariatric Surgery. Anesth Analg. 2019 Jul;129(1):51-60. doi: 10.1213/ANE.0000000000003696. PMID 30113392
- [Result] Amer MA, Smith MD, Herbison GP, Plank LD, McCall JL. Network meta-analysis of the effect of preoperative carbohydrate loading on recovery after elective surgery. Br J Surg. 2017 Feb;104(3):187-197. doi: 10.1002/bjs.10408. Epub 2016 Dec 21. PMID 28000931
- [Result] Thorell A, MacCormick AD, Awad S, Reynolds N, Roulin D, Demartines N, Vignaud M, Alvarez A, Singh PM, Lobo DN. Guidelines for Perioperative Care in Bariatric Surgery: Enhanced Recovery After Surgery (ERAS) Society Recommendations. World J Surg. 2016 Sep;40(9):2065-83. doi: 10.1007/s00268-016-3492-3. PMID 26943657